CLINICAL TRIAL: NCT04030780
Title: Effect of Spore-forming Probiotics in Functional Dyspepsia Patients: a Randomized Placebo-controlled Trial
Brief Title: Effect of Sporebiotics in FD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: MY HEALTH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S62043
Record Dates: First submitted 2019-06-03; First posted 2019-07-24 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2020-07

CONDITIONS: Dyspepsia; Dysbiosis
Keywords: spore-forming probiotic; sporebiotic; proton pump inhibitor; dyspepsia
MeSH Terms: conditions — Dyspepsia; Dysbiosis

STUDY DESIGN:
Intervention Model Description: randomized placebo-controlled study in 2 parallel FD cohorts
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: participants, care providers, investigators and outcomes assessor are blinded during the randomized placebo-controlled phase (8 weeks) but not during the open-label extension phase (8 weeks)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1FD (on-PPI+sporebiotics) (Active Comparator): study procedures at inclusion (1) and after 8 weeks on-PPI+ sporebiotics (2) followed by 8 weeks on-PPI+ sporebiotics (open label)
  Interventions: Dietary Supplement: spore-forming probiotic
- Cohort 1FD (on-PPI+placebo) (Placebo Comparator): study procedures at inclusion (1) and after 8 weeks on-PPI+ placebo (2) followed by 8 weeks on-PPI+ sporebiotics (open label)
  Interventions: Other: Placebo
- Cohort 2FD (off-PPI+sporebiotics) (Active Comparator): study procedures at inclusion (1) and after 8 weeks of sporebiotics (2) followed by 8 weeks of sporebiotics (open label)
  Interventions: Dietary Supplement: spore-forming probiotic
- Cohort 2FD (off-PPI+placebo) (Placebo Comparator): study procedures at inclusion (1) and after 8 weeks of placebo (2) followed by 8 weeks of sporebiotics (open label)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: spore-forming probiotic — spore-forming probiotic administered as 1 capsule twice daily (2,5 x 109 CFU per capsule) during 8 weeks
  Arms: Cohort 1FD (on-PPI+sporebiotics); Cohort 2FD (off-PPI+sporebiotics)
Other: Placebo — similar capsules administered twice daily
  Arms: Cohort 1FD (on-PPI+placebo); Cohort 2FD (off-PPI+placebo)

SUMMARY:
Single-site prospective interventional study aiming to demonstrate the effect of spore-forming probiotics on dyspeptic symptoms and blood, saliva and stool parameters in FD patients with and without acid suppression, compared to placebo.

DETAILED DESCRIPTION:
Prospective randomized placebo-controlled study in 2 parallel FD cohorts (8 weeks) with open-label extension phase (8 weeks):

* cohort 1FD (on-PPI): study procedures at inclusion (1) and after 8 weeks on-PPI+ sporebiotics or placebo (2) followed by 8 weeks on-PPI+ sporebiotics (open label)
* cohort 2FD (off-PPI): study procedures at inclusion (1) and after 8 weeks of sporebiotics or placebo (2) followed by 8 weeks of sporebiotics (open label)

Clinical outcomes and blood, saliva and stool parameters will be assessed at the beginning and end of each treatment period (week 0, 8 and 16) with additional questionnaires after 1 month (week 4 and 12).

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years with FD diagnosis (Rome IV criteria)
* Male or female (not pregnant or lactating and using contraception or postmenopausal)
* Normal bowel habits (defecation once every 3 days up to 3 times a day)
* Witnessed written informed consent
* Access to home freezer (-18 to -20°C)
* Capable to understand and comply with the study requirements

Exclusion Criteria:

* Any active somatic or psychiatric condition that may explain dyspeptic symptoms (stable dose of single antidepressant allowed for psychiatric indication, no limitation for other indications)
* Predominant symptoms of gastro-esophageal reflux disease (GERD) or irritable bowel syndrome (IBS)
* Use of immunosuppressants or antibiotics <3 months
* History of major abdominal surgery (except for appendectomy, cholecystectomy or splenectomy)
* Personal history of diabetes mellitus type 1, celiac disease or inflammatory bowel disease
* Diabetes mellitus type 2 (including therapy)
* Active malignancy (including therapy)
* Known HIV, HBV or HCV infection (including therapy)
* Significant alcohol use (>10 units/weeks)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of clinical responders (first 8 weeks) in sporebiotics vs. placebo | 8 weeks
  The Leuven Postprandial Distress Scale (LPDS) is a daily diary assessing the severity of 11 upper gastrointestinal symptoms scored from 0 (none) to 4 (very severe). A difference of 0.7 from baseline for the cardinal PDS symptoms (average of first 3 questions) will be used as a cut-off to determine clinical response by comparing averaged pre-treatment scores with the average score during the last week on treatment with sporebiotics vs. placebo. Only subjects with baseline score >1 (mild) will be included in the intention-to-treat and per-protocol analysis.

SECONDARY OUTCOMES:
Proportion of minimal clinical responders (first 8 weeks) in sporebiotics vs. placebo | 8 weeks
  The Leuven Postprandial Distress Scale (LPDS) is a daily diary assessing the severity of 11 upper gastrointestinal symptoms scored from 0 (none) to 4 (very severe). Proportion of minimal clinical responders using the minimum clinically important difference (MCID) of 0.5 for the cardinal PDS symptoms (first 3 questions) in subjects with baseline score >1 (mild) will be compared between sporebiotics and placebo for both cohorts combined.
Change in weekly PDS symptoms from baseline (first 8 weeks) on sporebiotics vs. placebo and changes within-groups | 8 weeks
  The Leuven Postprandial Distress Scale (LPDS) is a daily diary assessing the severity of 11 upper gastrointestinal symptoms scored from 0 (none) to 4 (very severe). Change in weekly PDS symptoms (first 3 questions) will be compared within- and between-treatments for both cohorts combined.
Change in weekly EPS symptoms from baseline (first 8 weeks) on sporebiotics vs. placebo and changes within-groups | 8 weeks
  The Leuven Postprandial Distress Scale (LPDS) is a daily diary assessing the severity of 11 upper gastrointestinal symptoms scored from 0 (none) to 4 (very severe). Change in weekly EPS symptoms (questions 4+5) will be compared within- and between-treatments for both cohorts combined.
Change in weekly individual symptoms from baseline (first 8 weeks) on sporebiotics vs. placebo and changes within-groups | 8 weeks
  The Leuven Postprandial Distress Scale (LPDS) is a daily diary assessing the severity of 11 upper gastrointestinal symptoms scored from 0 (none) to 4 (very severe). Change in weekly individual symptoms will be compared within- and between-treatments for both cohorts combined.
Proportion of (minimal) clinical responders (3 of the last 4 weeks of treatment) in sporebiotics vs. placebo | 8 weeks
  Proportion of (minimal) clinical responders for the cardinal PDS symptoms (first 3 questions) in subjects with baseline score >1 (mild) will be compared for 3 of the last 4 weeks of treatment between sporebiotics and placebo for both cohorts combined.
Weekly (minimal) clinical responder rates in sporebiotics vs. placebo | 8 weeks
  Change in weekly proportions for the cardinal PDS symptoms (first 3 questions) in subjects with baseline score >1 (mild) will be compared within- and between-treatments for both cohorts combined.
Change in monthly PAGI-SYM score from baseline (first 8 weeks) on sporebiotics vs. placebo and changes within-groups | 8 weeks
  The Patient Assessment of GastroIntestinal SYMptom severity (PAGI-SYM) is a validated questionnaire assessing the severity of 20 symptoms scored from 0 (none) to 4 (very severe). Change in monthly scores will be compared within- and between-treatments for both cohorts combined.
Change in monthly PAGI-QOL score from baseline (first 8 weeks) on sporebiotics vs. placebo and changes within-groups | 8 weeks
  The Patient Assessment of GastroIntestinal Quality Of Life (PAGI-QOL) is a validated questionnaire assessing 30 items scored from 0 (all the time) to 5 (none of the time). Change in monthly scores will be compared within- and between-treatments for both cohorts combined.
Change in high-sensitivity C-reactive protein (hs-CRP) on sporebiotics vs. placebo and changes within-groups | 8 weeks
  Change in hs-CRP (mg/L) sporebiotics vs. placebo and within-group by comparing pre- with post-treatment values.
Change in peripheral blood mononuclear cells on sporebiotics vs. placebo and changes within-groups | 8 weeks
  Change in proportion of PBMC (measured by flow-cytometry) on sporebiotics vs. placebo and changes within-groups by comparing pre- with post-treatment values.
Change in plasma cytokines on sporebiotics vs. placebo and changes within-groups | 8 weeks
  Change in cytokines (measured by multiplex) on sporebiotics vs. placebo and changes within-groups by comparing pre- with post-treatment values.
Change in lipopolysaccharide-binding protein (LBP) on sporebiotics vs. placebo and changes within-groups | 8 weeks
  Change in LBP (ng/mL) on sporebiotics vs. placebo and changes within-groups by comparing pre- with post-treatment values.
Change in stool microbiota on sporebiotics vs. placebo and changes within-groups | 8 weeks
  Change in stool microbiota (quantitative microbiota profiles) on sporebiotics vs. placebo and changes within-groups by comparing pre- with post-treatment values.
Safety of sporebiotics vs. placebo | 16 weeks
  number of adverse events with sporebiotics vs. placebo

CONTACTS AND LOCATIONS:
Overall Officials: Tim Vanuytsel, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wauters L, Slaets H, De Paepe K, Ceulemans M, Wetzels S, Geboers K, Toth J, Thys W, Dybajlo R, Walgraeve D, Biessen E, Verbeke K, Tack J, Van de Wiele T, Hellings N, Vanuytsel T. Efficacy and safety of spore-forming probiotics in the treatment of functional dyspepsia: a pilot randomised, double-blind, placebo-controlled trial. Lancet Gastroenterol Hepatol. 2021 Oct;6(10):784-792. doi: 10.1016/S2468-1253(21)00226-0. Epub 2021 Aug 3. PMID 34358486